CLINICAL TRIAL: NCT06210139
Title: Evaluating the Prescribing Pattern and Knowledge, Attitude and Practice as Well as the Adherence Level to Iron Chelation Therapy in Thalassemia
Brief Title: Pharmacotherapy Prescribing Pattern and the Adherence Level to Iron Chelation Therapy in Thalassemia
Status: Completed | Type: Observational
Sponsor: Reem Ali Shaker (Other)
Responsible Party: Sponsor-Investigator, Reem Ali Shaker, Principle investigator, Kufa University
Organization: Kufa University (Other)
Other Study IDs: MEC-40
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Thalassemia
Keywords: thalassemia; prescribing pattern; knowledge; adherence
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thalassemias are a heterogeneous grouping of genetic disorders that result in dysfunctional Hb, reduced RBC life span leading to chronic anemia . Thalassemia is endemic in the Middle East. Iron chelation therapy (ICT) is one of treatment used however ICT is associated with patients adherence problem thus impacting its effectiveness .

DETAILED DESCRIPTION:
Thalassemias are a heterogeneous grouping of genetic disorders that result from a decreased synthesis of alpha or beta chains of hemoglobin resulting in dysfunctional Hb, reduced RBC life span and hemolytic anemia as well as ineffective erythropoiesis leading to chronic anemia. Thalassemia is endemic in the Middle East, the Mediterranean region, and Southeast Asia, its prevalence in these region range from 7%-10%. There are 3 iron chelators licensed for clinical use, namely, deferoxamine (DFO), deferiprone (DFP), and deferasirox (DFX). Advancement in blood transfusions and ICT transforms this disease from fatal childhood disease to adult chronic disease . From other side, thalassemic patients on ICT suffering from therapy related challenge such as nonadherence, Nonadherence to ICT remains a long-standing and serious issue in thalassemia with ranges from 30% to 80% World widely. Issue of nonadherence and suboptimal responsiveness to ICT is complex and multifactorial such as side effects and administrations on top of inadequate knowledge and practice lead to reduced adherence to ICT thus increasing morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* male and female patients with age above 3 years old diagnosed with thalassemia,
* having iron overload
* taken Iron chelation therapy
* having the acceptance to participate in the study.

Exclusion Criteria:

* renal and hepatic impairment,
* Allergic to any drug of the study
* history of viral hepatitis or HIV
* Gastrointestinal disorder affecting drug absorption.
* psychiatric disorder affecting consent agreement and unable to comply with study.

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be conducted on the patients diagnosed with thalassemia and treated with iron chelation therapy who admitted to thalassemia center of AL Zahraa teaching hospital in AL Najaf Governorate-Iraq
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Adherence level | Baseline
  assessing patient adherence level to oral iron chelation therapy by Morisky medication adherence scale- 8 ( score less than 6 considered as low adherence , 6-7 medium adherence and 8 score considered as high adherence
KAP score | Baseline
  assessment of KAP( knowledge , attitude and practice) by using modified Bloom's cut-off value of 70% was used to classify patient's KAP into poor/negative for those with score below 70% and good/positive for those with score above 70%

SECONDARY OUTCOMES:
prescribing pattern | Baseline
  describe the pharmacotherapy prescribing pattern in thalassemia
Association of patient's factors with poor adherence | Baseline
  exploring the association between patient's factors with adherence level by multivariate analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fadhil A Riziji, PhD, Study Director — Kufa university/ faculty of pharmacy
Locations (1):
- AL Zahar teaching Hospital, Najaf, Iraq

IPD SHARING:
Plan to Share IPD: No